CLINICAL TRIAL: NCT03620305
Title: Septic Pseudarthrosis Of Long Bone : Experience In A Regional Reference Center
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Principal Investigator, Eugénie MABRUT, CRA, Hospices Civils de Lyon
Other Study IDs: 18-078
Record Dates: First submitted 2018-07-27; First posted 2018-08-08 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Pseudoarthrosis of Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Description of treatment of septic pseudarthrosis: chirurgical and medical treatment
  Interventions: Other: Description of treatment of septic pseudarthrosis

INTERVENTIONS:
Other: Description of treatment of septic pseudarthrosis — description of chirurgical 2 steps management of septic pseudarthrosis

SUMMARY:
Description of septic pseudarthrosis with chirurgical treatment in two steps (first step : Implementation of cement, second step : bone reconstruction, with or without device)

ELIGIBILITY:
Inclusion Criteria:

* patients having septic pseudarthrosis of long bone treated at the CRIOAc LYON

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: : patients having septic pseudarthrosis managed with 2 steps chirurgical treatment
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Description of treatment of septic pseudarthrosis : chirurgical treatment - rate of use of this type of chirurgical treatment among patients with septic pseudarthrosis | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Description of treatment of septic pseudarthrosis : chirurgical treatment

SECONDARY OUTCOMES:
Description of treatment of septic pseudarthrosis : medical treatment - duration of treatment in patients having sepstic pseudarthrosis | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Description of treatment of septic pseudarthrosis : medical treatment
Treatment failure : rate of failure with this 2 times chirurgical treatment | Outcome is measured at the end of follow-up (usually between 12 and 24 months after antibiotic therapy disruption)
  Treatment failure is defined by local clinical and/or microbiological relapse; and/or need for additional surgery; death of septic origin

CONTACTS AND LOCATIONS:
Overall Officials: Tristan Ferry, Principal Investigator — Hospices Civils de Lyon - Hôpital Croix-Rousse
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided